CLINICAL TRIAL: NCT01644201
Title: A Randomized, Double Blind, Placebo Controlled Trial Evaluating the Effects of a Highly Viscous Non-starch Polysaccharide (PolyGlycopleX® - PGX®), on Glycemic Control, Cardiometabolic Risk Factors and Weight Loss in Overweight and Obese Type II Diabetics Enrolled in a Medically Supervised Weight Management Program.
Brief Title: A Study Evaluating the Effects of a High Viscosity Non-starch Polysaccharide (PolyGlycopleX® - PGX®) on Glycemic Control, Cardiometabolic Risk Factors and Weight Loss in Overweight and Obese Type II Diabetics
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: Too slow recruitment
Sponsor: InovoBiologic Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: Wharton Study No. 05
Record Dates: First submitted 2012-07-16; First posted 2012-07-19 (Estimated); Last update posted 2021-02-11 (Actual); Status verified 2015-08

CONDITIONS: Type II Diabetes Mellitus; Obesity
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Obesity | interventions — PolyGlycoplex; Flour

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- High viscosity non-starch polysaccharide, PolyGlycopleX®-PGX® (Active Comparator)
  Interventions: Dietary Supplement: PolyGlycopleX® - PGX®
- Placebo (Rice Flour) (Placebo Comparator)
  Interventions: Dietary Supplement: Rice Flour (placebo)

INTERVENTIONS:
Dietary Supplement: PolyGlycopleX® - PGX® — 15g or 20g total daily dose, 5g pre-mixed with liquid meal replacement and consumed twice daily, 5g supplement granules sprinkled on food and consumed once of twice daily
  Arms: High viscosity non-starch polysaccharide, PolyGlycopleX®-PGX®
Dietary Supplement: Rice Flour (placebo) — 15g or 20g total daily dose, 5g pre-mixed with liquid meal replacement and consumed twice daily, 5g supplement granules sprinkled on food and consumed once of twice daily
  Arms: Placebo (Rice Flour)

SUMMARY:
One out of two adults in Canada is currently overweight and therefore at increased risk for a number of medical conditions including diabetes, high blood pressure, heart attacks and stroke. Obesity is less prevalent in populations consuming large amounts of dietary fibre, suggesting that fibre intake could play an important role in prevention and progression of obesity and diabetes and other conditions. Several studies have suggested that fibre has a positive effect on blood sugar and may help lower body weight.

The purpose of this study is to help better understand the effect of adding fibre supplementation to a low calorie diet on blood sugar control and weight loss. The investigators hypothesize that blood sugar control will improve in participants in the fibre supplementation group.

Men and women, with stable Type 2 Diabetes (e.g. no medication change in the last 3 months), between 18 - 75 years of age, and with a Body Mass Index (BMI) between 27 - 60 kg/m2 can participate in this study.

ELIGIBILITY:
Inclusion Criteria:

* 18-75 years of age (if >65 years of age, enrolment at the discretion of qualified investigator)
* BMI 27-60 Kg/m2
* Stable Type 2 diabetes mellitus (i.e. no medication change in the last 3 months)
* Ability to provide written informed consent in accordance with Good Clinical Practice (GCP) and local legislation

Exclusion Criteria:

* HbA1c <7.0% or >10.0%
* History of any bariatric surgery
* >10 Kg weight gain or weight loss in the past 3 months
* Known eating disorder
* Participant has taken weight loss medication in the last 3 months (eg. Meridia, Xenical)
* Participant is taking any of the following medications that can alter body weight or appetite:

  * Antipsychotics or neuroleptics
  * Prednisone
  * Antidepressants

    * Tricyclic such as amitriptyline, imipramine (Tofranil), and doxepin (Sinequan)
    * Monoamine oxidase inhibitors (MAOIs) such as tranylcypromine, (Parnate), isocarboxazid (Marplan) and phenelzine (Nardil)
    * Tetracyclic such as Mirtazapine (Remeron)
    * Serotonin antagonist and reuptake inhibitors (SARI) such as Trazodone

Note: The following antidepressants are NOT exclusion medications:

* SSRIs such as citalopram (Celexa), escitalopram (Lexapro), fluvoxamine (Luvox), fluoxetine (Prozac), sertraline (Zoloft), paroxetine (Paxil)
* Wellbutrin
* SNRIs such as venlafaxine (Effexor), duloxetine (Cymbalta)

  * Participant is taking any of the following natural health products that can alter body weight or appetite: ephedra, synephrine, green tea extracts, daily use of bulk fibre laxatives (e.g. psyllium, glucomannan)
  * Participant not eligible for enrolment in a medically supervised LCD program at the Wharton Medical Clinic (WMC only accepts patients by referral from a family physician. To be eligible patients must have a BMI ≥ 30 or ≥ 27 with at least one obesity related comorbidity.)
  * Patient with a past history of severe hypoglycaemia (as defined by the Diabetes Control and Complications Trial (DCCT)) whether or not on insulin, sulfonylureas and non-sulfonylurea secretogogues
  * Patient with documented hypoglycemic unawareness, whether or not on insulin, sulfonylureas and non-sulfonylurea secretogogues
  * Achalasia (i.e. difficulty swallowing)
  * Patient is taking medication that targets GLP-1 (glucagon-like peptide-1) including GLP-1 analogues (e.g. Byetta (Exenatide), Victoza (Liraglutide)) and DPP-IV inhibitors (e.g. Januvia(Sitagliptin), Onglyza (Saxagliptin).
  * Positive urine pregnancy test, pregnancy, breast feeding, or hormonal contraceptives started in the last 6 months prior to the start of the study
  * Absence of a highly effective method of birth control for female of childbearing potential (premenopausal or not surgically sterile) OR does not plan to use contraception for the duration of study participation AND does not agree to periodic urine pregnancy testing during the study. ICH M3 defines a highly effective method of birth control as those which result in a low failure rate (i.e. less than 1% per year) when used consistently and correctly such as implants, injectables, combined oral contraceptives, some IUDs, sexual abstinence or vasectomised partner.
  * Substance abuse: tobacco (including those who have quit smoking in the last 12 months), Cannabis sativa, or other controlled substances use
  * Any allergies to study product ingredients including dairy, whey, rice, soy and or coconut.
  * Labile or uncontrolled hypertension (SBP ≥ 160 mmHg and/or DBP ≥ 100 mmHg)
  * Current diagnosis or history of gastrointestinal diseases or disorders (with the exception of Irritable Bowel Syndrome and GERD at the discretion of qualified investigator).
  * Heart failure
  * Substantial neurological or psychological illness within the last 6 months (at the discretion of qualified investigator)
  * Contraindications to LCD

    1. any major surgery that is, at the time of screening, planned to take place during the study
    2. history of drug or alcohol dependency within six months prior to signing the informed consent form.
    3. history of active malignancy (exceptions at the discretion of qualified investigator e.g. squamous cell carcinoma), chronic inflammatory disorder, or chronic infections which would interfere with protocol completion
    4. history of CV event or angina within 6 months (with the exception of stable angina at the discretion of qualified investigator)
    5. history of active gall bladder disease where the gallbladder was not removed
    6. inflammatory bowel disease
    7. type 1 diabetes
    8. significant renal impairment eGFR < 50
    9. porphyria
    10. cirrhosis
    11. patients deemed unable to comprehend or comply with the diet and/or,
    12. unable to attend program follow up visits
  * Participant cannot fully understand all instructions in English.
  * Any other medical, social or geographic condition, which, in the opinion of the qualified investigator would not allow safe completion of the protocol.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Actual)
Dates: Start 2012-10; Primary Completion 2016-11 (Actual); Study Completion 2016-11 (Actual)

PRIMARY OUTCOMES:
HbA1c | End of study (1 year)

CONTACTS AND LOCATIONS:
Overall Officials: Sean Wharton, MD, FRCPC, PharmD, Principal Investigator
Locations (1):
- Wharton Medical Clinic and Weight Management Centre, Hamilton, Ontario, Canada

REFERENCES:
- [Derived] Reimer RA, Wharton S, Green TJ, Manjoo P, Ramay HR, Lyon MR, Gahler RJ, Wood S. Effect of a functional fibre supplement on glycemic control when added to a year-long medically supervised weight management program in adults with type 2 diabetes. Eur J Nutr. 2021 Apr;60(3):1237-1251. doi: 10.1007/s00394-020-02328-8. Epub 2020 Jul 8. PMID 32642971